CLINICAL TRIAL: NCT06386887
Title: The Feasibility, Safety, and Clinical Outcomes of Fasting During Neoadjuvant Chemotherapy in Patients With Epithelial Ovarian Cancer
Brief Title: Fasting During Neoadjuvant Chemotherapy in Patient With Epithelial Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE1824
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Short term fasting; Intermittent fasting; Intermittent energy restriction (IER); Fasting mimicking diet (FMD)
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Intermittent Fasting | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Two arm, randomized, controlled study.
Who Masked: Outcomes Assessor
Masking Description: Participants' cross-sectional skeletal muscle areas will be measured. Measurements will be performed on CT scans obtained within 4-6 weeks of treatment initiation (with a 7-day screening window) by a fellowship-trained, experienced radiologist and imaging specialist in consensus who will be blinded to participant clinical variables and treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting (Experimental): Participants will receive 16 hours of fasting, 8 hour regular feeding for 5 days a week starting 2 days prior to chemotherapy.
  Interventions: Behavioral: Intermittent Fasting; Drug: Neoadjuvant chemotherapy
- Standard of Care (Active Comparator): Participants will receive standard of care dietary recommendations and will provide a 3-day diet diary at study enrollment and during cycles 2 and 3.
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Behavioral: Intermittent Fasting — Intermittent fasting (IF) also known as time restricted eating regimen consisting of 16 hours of fasting and 8 hours of ad libitum feeding for 5 days followed by ad libitum feeding for 2 days has been proposed. With this type of intervention, there are no dietary restrictions to the type or quality of food and it decreased daily energy intake by 20%. Participants will be asked to follow an IF schedule consisting of 16 hour of continuous fasting per day for 5 days a week. This will be started 2 days prior to chemotherapy (cycle 2).
  Other Names: Time restricted eating
  Arms: Intermittent Fasting
Drug: Neoadjuvant chemotherapy — Chemotherapy will be given as standard treatment every 3 weeks (21 days) and continue for 3 to 4 cycles per routine care. As chemotherapy is not part of this research study, participants will begin standard chemotherapy as decided by their physician.

SUMMARY:
The goal of this clinical trial is to see if timed fasting (periods of time that you don't eat) in participants who are receiving chemotherapy prior to surgery is achievable, safe and can improve quality of life, symptoms and outcomes (results) compared to participants who receive standard dietary recommendations in individuals being treated for epithelial ovarian cancer . The main questions it aims to answer are:

* Is it feasible to use intermittent fasting during neoadjuvant chemotherapy?
* Is it safe to use intermittent fasting during neoadjuvant chemotherapy?
* Do participants find it acceptable to use intermittent fasting during neoadjuvant chemotherapy?

Researchers will compare participants who receive standard dietary recommendations to see which method is more achievable, safe, and able to improve quality of life, symptoms and outcomes.

Participants will:

* Receive either the fasting intervention (schedule of times when you do not eat) or standard diet recommendations for 6-9 weeks prior to your surgery starting with the second cycle of chemotherapy.
* All participants will be asked to complete chemotherapy and surgery, cancer imaging, baseline screening tests, nutritional assessments, food diaries, blood tests, and surveys about wellbeing.
* Participants in the intervention group will be asked to follow a fasting schedule that consists of not eating for 16 hours a day followed by normal eating for the remaining 8 hours of the day for 5 days in a row followed by 2 days of regular eating each week.

DETAILED DESCRIPTION:
The quality of diet can affect the biology of cancer. For example, evidence implies a high fat/ Western diet may impose adverse events on ovarian cancer outcomes, and the potential that the gut microbiome alterations secondary to dietary changes may impact tumor responsiveness to treatment and outcomes. This study seeks to clarify the effect of dietary intervention on the tumor and gut microbiome and ovarian cancer biology. The objectives of this study include:

* Primary: To test the feasibility and safety of IF during neoadjuvant chemotherapy (including effects on body composition)
* Secondary: To measure the effects of IF on participant reported outcomes, chemotherapy toxicity and quality of life.
* Exploratory: To test the effect of IF on pathologic response, systemic inflammatory and immune responses, microbial diversity and metabolic pathway alterations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Participants with confirmed diagnosis of primary epithelial ovarian cancer (EOC) by internal cytologic or histologic evaluation (including fallopian tube and primary peritoneal cancer)
* Participants receiving platinum-based chemotherapy for ovarian cancer including

  * Participants with stage III or IV EOC planned to undergo neoadjuvant chemotherapy (including participants who had a diagnostic laparoscopy or aborted debulking) OR
  * Participants with stage III or IV EOC following primary debulking surgery
  * Participants with recurrent epithelial ovarian cancer who will receive platinum-based chemotherapy OR
  * Participants who had undergone neoadjuvant chemotherapy and interval debulking surgery who will be receiving adjuvant (postoperative) chemotherapy
* Any invasive ovarian cancer histology
* Normal cognitive function

Exclusion Criteria:

* Age <18 years
* Malignant complete or partial bowel obstruction confirmed on imaging.
* Participants unable to provide informed consent.
* BMI <18
* Participants diagnosed with severe malnutrition as assessed by study dietitian
* Type I diabetes on insulin
* Absence of pretreatment CT abdomen and pelvis imaging or >4-6 weeks between imaging and cycle 1 of chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Intermittent fasting compliance as measured by serum glucose laboratory testing | Day 1 of cycle 1 (each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (serum glucose) prior to each chemotherapy.
Intermittent fasting compliance as measured by ketone laboratory testing | Day 1 of cycle 1 (each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (ketone) prior to each chemotherapy.
Intermittent fasting compliance as measured by IGF-1 laboratory testing | Day 1 of cycle 1 (each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (IGF-1) prior to each chemotherapy.
Intermittent fasting compliance as measured by insulin laboratory testing | Day 1 of cycle 1 (each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (insulin) prior to each chemotherapy.
Intermittent fasting compliance as measured by serum glucose laboratory testing | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (serum glucose) prior to each chemotherapy.
Intermittent fasting compliance as measured by ketone laboratory testing | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (ketone) prior to each chemotherapy. which will be measured by metabolic laboratory tests (serum glucose, ketone, IGF-1, and insulin) prior to each chemotherapy.
Intermittent fasting compliance as measured by IGF-1 laboratory testing | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (IGF-1) prior to each chemotherapy.
Intermittent fasting compliance as measured by insulin laboratory testing | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (insulin) prior to each chemotherapy.
Intermittent fasting compliance as measured by serum glucose laboratory testing | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (serum glucose) prior to each chemotherapy.
Intermittent fasting compliance as measured by ketone laboratory testing | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (ketone) prior to each chemotherapy.
Intermittent fasting compliance as measured by IGF-1 laboratory testing | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (IGF-1) prior to each chemotherapy.
Intermittent fasting compliance as measured by insulin laboratory testing | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by metabolic laboratory tests (insulin) prior to each chemotherapy.
Intermittent fasting compliance as measured by self-reported assessment | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by a self-reported compliance checklist assessment.
Intermittent fasting compliance as measured by self-reported assessment | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured by a self-reported compliance checklist assessment.
Intermittent fasting compliance as measured by food diary | Week 3 (Day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured a 3-food diary submitted during each dietitian in person visit.
Intermittent fasting compliance as measured by food diary | Week 6 (Day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will be assessed for intermittent fasting compliance which will be measured a 3-food diary submitted during each dietitian in person visit.
Intermittent fasting compliance as measured by food diary | Up to 12 weeks post intervention
  Participants will be assessed for intermittent fasting compliance which will be measured a 3-food diary submitted during each dietitian in person visit.
Pre body composition | Baseline
  Pre- and post- treatment body composition will be assessed by Computed Tomography scans.
Post body composition | Up to 12 weeks post intervention
  Pre- and post- treatment body composition will be assessed by Computed Tomography scans.

SECONDARY OUTCOMES:
Chemotherapy related toxicity at Cycle 2 | Week 3 (At day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will undergo evaluation of chemotherapy related toxicity (according to Common Terminology Criteria for Adverse Events [CTCAE version 5.0]).
Chemotherapy related toxicity at Cycle 3 | Week 6 (At day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will undergo evaluation of chemotherapy related toxicity (according to Common Terminology Criteria for Adverse Events [CTCAE version 5.0]).
Chemotherapy related toxicity at Cycle 4 | Week 9 (At day 1 of cycle 4; each cycle consisting of 21 days)
  Participants that undergo an additional cycle of chemotherapy will undergo evaluation of chemotherapy related toxicity (according to Common Terminology Criteria for Adverse Events [CTCAE version 5.0]).
Chemotherapy related toxicity at post treatment | Up to 12 weeks post intervention
  Participants will undergo evaluation of chemotherapy related toxicity (according to Common Terminology Criteria for Adverse Events [CTCAE version 5.0]),
ESAS Score at Enrollment | At baseline
  Participants will complete Edmonton Symptom Assessment Questionnaires (ESAS) at enrollment. The ESAS assesses pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
ESAS Score at Cycle 2 | Week 3 (At day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will complete Edmonton Symptom Assessment Questionnaires (ESAS). The ESAS assesses pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
ESAS Score at Cycle 3 | Week 6 (At day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will complete Edmonton Symptom Assessment Questionnaires (ESAS). The ESAS assesses pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
ESAS Score at Post Treatment | Up to 12 weeks post intervention
  Participants will complete Edmonton Symptom Assessment Questionnaires (ESAS). The ESAS assesses pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
SF-125 Score at Baseline | At baseline
  Participants will complete Study Short Form-12 Health Survey (SF-125) at enrollment. The SF-12 measures physical and mental health status. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
SF-125 Score at Cycle 2 | Week 3 (At day 1 of cycle 2; each cycle consisting of 21 days)
  Participants will complete Study Short Form-12 Health Survey (SF-125) day 1 cycle 2. The SF-12 measures physical and mental health status. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
SF-125 Score at Cycle 3 | Week 6 (At day 1 of cycle 3; each cycle consisting of 21 days)
  Participants will complete Study Short Form-12 Health Survey (SF-125) day 1 cycle 3. The SF-12 measures physical and mental health status. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
SF-125 Score at Post Treatment | Up to 12 weeks post intervention
  Participants will complete Study Short Form-12 Health Survey (SF-125) post treatment. The SF-12 measures physical and mental health status. Responses are scored to produce a physical component summary and a mental component summary on a scale from 0 to 100, with higher scores indicative of better functional status.
Pre Quality of Life (QLQ-C30) Score at Baseline | At baseline
  Quality of life questionnaires will be distributed at enrollment and will be compared between IF and control groups. Quality of life will be measured by Quality of life will be measured with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30). EORTC QLQ-C30 is a 30 item questionnaire. Higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Post Quality of Life (QLQ-C30) Score Post Treatment | Up to 12 weeks post intervention
  Quality of life questionnaires will be distributed at enrollment and will be compared between IF and control groups. Quality of life will be measured by Quality of life will be measured with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30). EORTC QLQ-C30 is a 30 item questionnaire. Higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Pre Functional Assessment (FACT-O) Score at Baseline | Up to 12 weeks post intervention
  Functional Assessment of Cancer Therapy- Ovarian (FACT-O) will be administered post treatment and will be compared between IF and control groups. FACT-O is a 39 item questionnaire with a 5 point Likert-type scale. Scores range from 0-156. The higher the score, the better the quality of life.
Post Functional Assessment (FACT-O) Score Post Treatment | Up to 12 weeks post intervention
  Functional Assessment of Cancer Therapy- Ovarian (FACT-O) will be administered at enrollment and will be compared between IF and control groups. FACT-O is a 39 item questionnaire with a 5 point Likert-type scale. Scores range from 0-156. The higher the score, the better the quality of life.
AIM Survey Score at Cycle 2 | Week 3 (At day 1 of cycle 2; each cycle consisting of 21 days)
  Acceptability of intervention Measure (AIM) questionnaire will be administered IF participants. AIM has 4 item psychometric assessment times measuring acceptability of intervention. Scale values range from 1 to 5. Overall scores that are lower indicating lower acceptability, and higher scores indicating greater acceptability, appropriateness, and feasibility.
AIM Survey Score at Cycle 3 | Week 6 (At day 1 of cycle 3; each cycle consisting of 21 days)
  Acceptability of intervention Measure (AIM) questionnaire will be administered IF participants. AIM has 4 item psychometric assessment times measuring acceptability of intervention. Scale values range from 1 to 5. Overall scores that are lower indicating lower acceptability, and higher scores indicating greater acceptability, appropriateness, and feasibility.
AIM Survey Score at Post Treatment | Up to 12 weeks post intervention
  Acceptability of intervention Measure (AIM) questionnaire will be administered IF participants. AIM has 4 item psychometric assessment times measuring acceptability of intervention. Scale values range from 1 to 5. Overall scores that are lower indicating lower acceptability, and higher scores indicating greater acceptability, appropriateness, and feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kuznicki, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Department of Subspecialty Care for Women's Health Women's Health; Division of Gynecologic Oncology, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected participant data will be shared through publication including clinical data, laboratory results, CT data, qualitative data (questionnaire's) in additional, molecular data, histologic data, treatment response after statistical analysis. All data will be shared without participant identifiers.
Time Frame: Anticipated 6-2025 - indefinitely through publication of data